CLINICAL TRIAL: NCT01617187
Title: A Multicenter, Randomized, Double-Blind, Fixed-Dose, 6-Week Trial of the Efficacy and Safety of Asenapine Compared With Placebo Using Olanzapine as an Active Control in Subjects With an Acute Exacerbation of Schizophrenia
Brief Title: A Study of the Efficacy and Safety of Asenapine in Participants With an Acute Exacerbation of Schizophrenia (P05688)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05688; 2010-018407-28 (EudraCT Number)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Asenapine 2.5 mg BID (Experimental)
  Interventions: Drug: Asenapine; Drug: Placebo Olanzapine
- Asenapine 5 mg BID (Experimental)
  Interventions: Drug: Asenapine; Drug: Placebo Olanzapine
- Olanzapine 15 mg QD (Active Comparator)
  Interventions: Drug: Placebo Asenapine; Drug: Olanzapine; Drug: Placebo Olanzapine
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo Asenapine; Drug: Placebo Olanzapine

INTERVENTIONS:
Drug: Asenapine — 2.5 mg or 5 mg fast dissolving active asenapine tablets administered sublingually
  Arms: Asenapine 2.5 mg BID; Asenapine 5 mg BID
Drug: Placebo Asenapine — Fast dissolving placebo asenapine tablets (to match 2.5 mg and 5 mg active asenapine tablets) administered sublingually
  Arms: Olanzapine 15 mg QD; Placebo BID
Drug: Olanzapine — 5 and 10 mg film-coated active olanzapine tablets administered orally QD. The time of the active olanzapine dose (either morning or evening) is not disclosed in order to preserve blinding
  Arms: Olanzapine 15 mg QD
Drug: Placebo Olanzapine — Film-coated placebo olanzapine tablets (to match 5 and 10 mg active olanzapine tablets) administered orally

SUMMARY:
The purpose of this trial is to assess the effect of asenapine 2.5 and 5 mg sublingually twice daily (BID) compared with placebo in the treatment of schizophrenia (overall symptoms) as measured by the Positive and Negative Syndrome Scale (PANSS). Olanzapine administered 15 mg orally once daily (QD) was used as an active control. The primary hypothesis is that at least one of the asenapine doses is superior to placebo in improving schizophrenia symptoms as measured by the change from Baseline in the PANSS total score at Day 42. The first key secondary hypothesis is that at least one of the asenapine doses is superior to placebo in improving schizophrenia symptoms as measured by the change from Baseline in Clinical Global Impression Scale-Severity (CGI-S) score at Day 42. The second key secondary hypothesis is that at least one of the asenapine doses is superior to placebo in improving schizophrenia symptoms as measured by the rate of PANSS responders (≥30% Reduction From Baseline in PANSS Total Score) at Day 42.

DETAILED DESCRIPTION:
The trial consists of a screening/tapering period, treatment period, and follow-up period. The 6-week active treatment period includes an inpatient phase and outpatient phase. Participants who complete the trial may continue treatment under a long-term extension protocol (P05689). Participants who do not continue in the treatment continuation trial (whether they complete the 6-week trial or discontinue prematurely) will have a follow-up visit 7 days after their last dose of trial medication.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of schizophrenia of paranoid, disorganized, or undifferentiated subtype
* Minimum PANSS total score of 70 at Screening and Baseline
* Score of at least 4 (moderate) in two or more of the five items in the positive subscale of the PANSS
* Confirmed to be experiencing an acute exacerbation of schizophrenia
* CGI-S scale score of at least 4 (moderately ill) at Baseline
* Has responded positively to an antipsychotic medication other than clozapine (Clozaril®) in a prior episode

Exclusion Criteria:

* Body mass index (BMI) <18.5 or >40.0 kg/m^2
* Laboratory and/or clinical evidence of clinically significant hepatic conditions
* Known history of, or undergoing treatment for, narrow angle glaucoma
* Diagnosed with epilepsy or has had any seizure disorder beyond childhood febrile seizures
* Known serological evidence of human immunodeficiency virus (HIV) antibody
* History of neuroleptic malignant syndrome or tardive dyskinesias
* Past or current diagnosis of schizoaffective disorder, schizophrenia of residual subtype, schizophrenia of catatonic subtype, current diagnosis of schizophrenia with course specifiers continuous, single episode in partial remission, or single episode in full remission, or borderline personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2014-08-11 (Actual); Study Completion 2014-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Landbloom R, Mackle M, Wu X, Kelly L, Snow-Adami L, McIntyre RS, Mathews M, Hundt C. Asenapine for the treatment of adults with an acute exacerbation of schizophrenia: results from a randomized, double-blind, fixed-dose, placebo-controlled trial with olanzapine as an active control. CNS Spectr. 2017 Aug;22(4):333-341. doi: 10.1017/S1092852916000377. Epub 2016 Nov 8. PMID 27821210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant randomized to asenapine 2.5 mg BID did not receive study drug but was recorded in clinical database as completing the study. In Participant Flow table, this participant is presented as Not Completed in period "Randomization through Start Treatment" (Not Treated).
Groups:
- Asenapine 2.5 mg BID: Participants were administered one 2.5 mg asenapine tablet twice daily (BID) for 42 days
- Asenapine 5 mg BID: Participants were administered one 5 mg asenapine tablet BID for 42 days
- Olanzapine 15 mg QD: Participants were administered 15 mg olanzapine (as one 10 mg and one 5 mg tablet) once daily (QD) for 42 days, except during Week 1 olanzapine 10 mg QD was administered
- Placebo BID: Participants were administered placebo tablets BID for 42 days
Period: Randomization Through Start Treatment
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Started | 98 (Randomized) | 113 (Randomized) | 46 (Randomized) | 103 (Randomized)
Completed | 97 | 113 | 46 | 101
Not Completed | 1 | 0 | 0 | 2
Not completed — Not Treated: Administrative Reason | 0 | 0 | 0 | 1
Not completed — Not Treated: Adverse Event | 0 | 0 | 0 | 1
Not completed — Not Treated: Completed study in database | 1 | 0 | 0 | 0
Period: Treatment Through Study Completion
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Started | 97 (Treated) | 113 (Treated) | 46 (Treated) | 101 (Treated)
Completed | 86 (Excludes the participant who did not receive study drug but completed study in database) | 102 | 41 | 91
Not Completed | 11 | 11 | 5 | 10
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 4 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 5 | 8 | 3 | 6
Not completed — Protocol Violation | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received ≥1 dose of study drug.
Groups:
- Asenapine 2.5 mg BID: Participants were administered one 2.5 mg asenapine tablet BID for 42 days
- Olanzapine 15 mg QD: Participants were administered 15 mg olanzapine (as one 10 mg and one 5 mg tablet) QD for 42 days, except during Week 1 olanzapine 10 mg QD was administered
- Total: Total of all reporting groups
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID | Total
Number analyzed (Participants) | 97 | 113 | 46 | 101 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.79) | 39.1 (10.68) | 40.8 (11.15) | 41.4 (12.05) | 40.6 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 44 | 18 | 47 | 148
  Male | 58 | 69 | 28 | 54 | 209
Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score (30 items) ranged from 30 to 210 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (Full Analysis Set [FAS]): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 93.3 (11.10) | 95.8 (13.77) | 92.7 (10.47) | 93.4 (11.16) | 94.1 (11.97)
Clinical Global Impression Scale-Severity (CGI-S) score [Mean (Standard Deviation); unit: score on a scale] — CGI-S is a 7-point scale for assessing the global severity of the participant's illness, with ratings from 1=normal, not ill to 7=very severely ill. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 4.8 (0.64) | 4.9 (0.64) | 4.8 (0.61) | 4.8 (0.61) | 4.8 (0.63)
Body Weight [Mean (Standard Deviation); unit: kg] | 81.6 (17.73) | 78.6 (17.88) | 80.7 (17.79) | 77.1 (17.56) | 79.3 (17.75)
PANSS negative subscale score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS negative subscale score (7 PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 23.5 (4.47) | 24.1 (4.50) | 23.4 (3.96) | 23.9 (4.22) | 23.8 (4.34)
PANSS positive subscale score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS positive subscale score (7 PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 24.4 (4.05) | 25.5 (4.76) | 24.6 (3.46) | 24.6 (3.88) | 24.8 (4.19)
PANSS general psychopathology subscale score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS general psychopathology subscale score (16 PANSS items) ranged from 16 to 112 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 45.5 (6.05) | 46.3 (6.87) | 44.7 (6.20) | 44.9 (6.05) | 45.5 (6.34)
PANSS Marder factor positive symptom score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder factor positive symptom score (calculated from value of 8 identified PANSS items) ranged from 8 to 56 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 29.3 (5.02) | 30.0 (5.05) | 29.0 (4.69) | 29.4 (4.36) | 29.5 (4.80)
PANSS Marder factor negative symptom score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder factor negative symptom score (calculated from value of 7 identified PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 22.6 (4.30) | 23.0 (4.66) | 23.0 (4.44) | 22.8 (4.76) | 22.8 (4.55)
PANSS Marder factor disorganized thought symptom score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder factor disorganized thought symptom score (calculated from value of 7 identified PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 21.5 (4.32) | 22.6 (4.93) | 21.2 (4.29) | 21.6 (4.42) | 21.8 (4.56)
PANSS Marder factor hostility/excitement symptom score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder factor hostility/excitement symptom score (calculated from value of 4 identified PANSS items) ranged from 4 to 28 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 9.0 (2.99) | 9.4 (3.49) | 8.7 (3.11) | 8.8 (3.22) | 9.0 (3.23)
PANSS Marder factor anxiety/depression symptom score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder factor anxiety/depression symptom score (calculated from value of 4 identified PANSS items) ranged from 4 to 28 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=96, 111, 45, 99 and 351 for asenapine 2.5 mg BID, asenapine 5 mg BID, olanzapine 15 mg QD, placebo BID and Total groups, respectively.
  score on a scale | 11.0 (2.97) | 10.9 (3.13) | 10.9 (3.62) | 10.7 (2.96) | 10.9 (3.09)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PANSS Total Score at Day 42
Description: The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 42; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 42
Population: FAS, defined as randomized participants who received ≥1 dose of study drug and had both a baseline and ≥1 post-baseline PANSS Total Score
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale | -17.4 (1.80) | -21.7 (1.60) | -21.6 (2.32) | -16.2 (1.71)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.6043, Mixed Model Repeated Measures (MMRM) — Adjusted p-value from graphical approach to control Type 1 error rate among primary and secondary efficacy hypotheses; Least Squares (LS) means difference = -1.3, 95% CI 2-sided [-6.1 to 3.6], Standard Error of Mean 2.46 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0356, MMRM — Adjusted p-value from graphical approach to control Type 1 error rate among primary and secondary efficacy hypotheses; LS means difference = -5.5, 95% CI 2-sided [-10.1 to -1.0], Standard Error of Mean 2.32 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Test type: Superiority or Other; p = 0.0587, MMRM — Unadjusted p-value; LS means difference = -5.4, 95% CI 2-sided [-11.1 to 0.2], Standard Error of Mean 2.86 — Olanzapine 15 mg BID minus Placebo BID

2. Secondary Outcome: Change From Baseline in CGI-S Score at Day 42
Description: Change from baseline in CGI-S score at Day 42 is a Key Secondary Outcome Measure. CGI-S is a 7-point scale for assessing the global severity of the participant's illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 42; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale | -0.9 (0.11) | -1.2 (0.10) | -1.1 (0.14) | -1.0 (0.11)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Confirmative testing of asenapine versus placebo for this measure was to be performed only if both asenapine doses were statistically superior to placebo in reduction from baseline in PANSS Total Score (Primary outcome measure); Test type: Superiority or Other; p = 0.9083, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.15 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0601, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.14 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Test type: Superiority or Other; p = 0.3898, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.18 — Olanzapine 15 mg BID minus Placebo BID

3. Secondary Outcome: Percentage of Participants Who Are PANSS Responders (≥30% Reduction From Baseline in PANSS Total Score) at Day 42
Description: Rate of PANSS responders at Day 42 is a Key Secondary Outcome Measure. A PANSS responder was defined as a participant who had a reduction from baseline of at least 30% in the PANSS total score at a post-baseline assessment. The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The Total score is the sum of the ratings for the individual items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. Missing data were imputed by Last Observation Carried Forward (LOCF).
Time Frame: Baseline and Day 42
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
percentage of participants | 14.6 (0.11) | 25.2 (0.10) | 26.7 (0.14) | 19.2 (0.11)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3700, Cochran-Mantel-Haenszel — P-value from Cochran Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1708, Cochran-Mantel-Haenszel — P-value from Cochran Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Test type: Superiority or Other; p = 0.2620, Cochran-Mantel-Haenszel — P-value from Cochran Mantel-Haenszel test with an adjustment for pooled center

4. Secondary Outcome: Change From Baseline in Body Weight at Day 42
Description: Change from baseline in body weight at Day 42 is the Key Safety Outcome Measure.
Time Frame: Baseline and Day 42
Population: All randomized participants who received ≥1 dose of study drug
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 97 | 113 | 46 | 101
kg | 1.3 (0.38) | 1.3 (0.33) | 2.4 (0.47) | 0.3 (0.35)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Olanzapine 15 mg QD; Test type: Superiority or Other; p = 0.0491, MMRM — p-value adjusted for multiple comparisons using Hochberg's method; LS means difference = -1.2, 95% CI 2-sided [-2.4 to -0.0], Standard Error of Mean 0.60 — Asenapine 2.5 mg BID minus Olanzapine 15 mg QD
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Olanzapine 15 mg QD; Test type: Superiority or Other; p = 0.0491, MMRM — p-value adjusted for multiple comparisons using Hochberg's method; LS means difference = -1.2, 95% CI 2-sided [-2.3 to -0.0], Standard Error of Mean 0.57 — Asenapine 5 mg BID minus Olanzapine 15 mg QD
Statistical Analysis 3: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0567, MMRM — Unadjusted p-value; LS means difference = 1.0, 95% CI 2-sided [-0.0 to 2.0], Standard Error of Mean 0.51 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 5 mg BID vs Placebo BID; Test type: Superiority or Other; p = 0.0391, MMRM — Unadjusted p-value; LS means difference = 1.0, 95% CI 2-sided [0.0 to 1.9], Standard Error of Mean 0.48 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Olanzapine 15 mg QD vs Placebo BID; Test type: Superiority or Other; p = 0.0003, MMRM — Unadjusted p-value; LS means difference = 2.2, 95% CI 2-sided [1.0 to 3.3], Standard Error of Mean 0.58 — Olanzapine 15 mg BID minus Placebo BID

5. Secondary Outcome: Change From Baseline in PANSS Total Score at Days 4, 7, 14, 21, 28 and 35
Description: The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28 and 35
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -4.0 (0.80) | -4.9 (0.76) | -5.5 (1.15) | -4.8 (0.81)
  Day 7 | -7.2 (1.17) | -9.1 (1.09) | -9.3 (1.67) | -7.1 (1.16)
  Day 14 | -9.9 (1.31) | -12.5 (1.19) | -12.4 (1.80) | -10.7 (1.28)
  Day 21 | -12.0 (1.55) | -14.8 (1.40) | -15.2 (2.09) | -13.2 (1.50)
  Day 28 | -12.3 (1.69) | -17.1 (1.49) | -17.3 (2.21) | -15.5 (1.61)
  Day 35 | -17.0 (1.66) | -19.0 (1.48) | -20.3 (2.19) | -15.4 (1.58)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.4849, MMRM — Unadjusted p-value; LS means difference = 0.8, 95% CI 2-sided [-1.4 to 2.9], Standard Error of Mean 1.09 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.8902, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-2.2 to 1.9], Standard Error of Mean 1.06 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.5826, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-3.4 to 1.9], Standard Error of Mean 1.36 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.9271, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-3.3 to 3.0], Standard Error of Mean 1.61 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1902, MMRM — Unadjusted p-value; LS means difference = -2.0, 95% CI 2-sided [-5.1 to 1.0], Standard Error of Mean 1.56 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.2710, MMRM — Unadjusted p-value; LS means difference = -2.2, 95% CI 2-sided [-6.2 to 1.7], Standard Error of Mean 2.00 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6773, MMRM — Unadjusted p-value; LS means difference = 0.7, 95% CI 2-sided [-2.8 to 4.3], Standard Error of Mean 1.79 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2895, MMRM — Unadjusted p-value; LS means difference = -1.8, 95% CI 2-sided [-5.2 to 1.6], Standard Error of Mean 1.72 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.4261, MMRM — Unadjusted p-value; LS means difference = -1.7, 95% CI 2-sided [-6.0 to 2.6], Standard Error of Mean 2.18 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5505, MMRM — Unadjusted p-value; LS means difference = 1.3, 95% CI 2-sided [-2.9 to 5.5], Standard Error of Mean 2.13 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4286, MMRM — Unadjusted p-value; LS means difference = -1.6, 95% CI 2-sided [-5.6 to 2.4], Standard Error of Mean 2.03 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4423, MMRM — Unadjusted p-value; LS means difference = -2.0, 95% CI 2-sided [-7.0 to 3.1], Standard Error of Mean 2.56 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.1691, MMRM — Unadjusted p-value; LS means difference = 3.2, 95% CI 2-sided [-1.4 to 7.7], Standard Error of Mean 2.30 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4682, MMRM — Unadjusted p-value; LS means difference = -1.6, 95% CI 2-sided [-5.8 to 2.7], Standard Error of Mean 2.17 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4961, MMRM — Unadjusted p-value; LS means difference = -1.8, 95% CI 2-sided [-7.2 to 3.5], Standard Error of Mean 2.71 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.4697, MMRM — Unadjusted p-value; LS means difference = -1.6, 95% CI 2-sided [-6.1 to 2.8], Standard Error of Mean 2.26 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0947, MMRM — Unadjusted p-value; LS means difference = -3.6, 95% CI 2-sided [-7.8 to 0.6], Standard Error of Mean 2.14 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0675, MMRM — Unadjusted p-value; LS means difference = -4.9, 95% CI 2-sided [-10.2 to 0.4], Standard Error of Mean 2.68 — Olanzapine 15 mg BID minus Placebo BID

6. Secondary Outcome: Percentage of Participants Who Are PANSS Responders (≥30% Reduction From Baseline in PANSS Total Score) at Days 4, 7, 14, 21, 28 and 35
Description: A PANSS responder was defined as a participant who had a reduction from baseline of at least 30% in the PANSS total score at a post-baseline assessment. The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The Total score is the sum of the ratings for the individual items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. Missing data were imputed by LOCF.
Time Frame: Days 4, 7, 14, 21, 28 and 35
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
percentage of participants
  Day 4 (n = 95,108,44,97) | 0.0 (0.27) | 0.0 (0.25) | 0.0 (0.38) | 2.1 (0.27)
  Day 7 (n = 96,111,45,99) | 2.1 (0.30) | 5.4 (0.28) | 0.0 (0.43) | 5.1 (0.30)
  Day 14 (n = 96,111,45,99) | 5.2 (0.31) | 5.4 (0.28) | 4.4 (0.42) | 7.1 (0.30)
  Day 21 (n = 96,111,45,99) | 8.3 (0.32) | 14.4 (0.29) | 11.1 (0.42) | 13.1 (0.31)
  Day 28 (n = 96,111,45,99) | 10.4 (0.36) | 16.2 (0.32) | 15.6 (0.47) | 14.1 (0.35)
  Day 35 (n = 96,111,45,99) | 15.6 (0.34) | 21.6 (0.30) | 15.6 (0.44) | 17.2 (0.32)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.1736, Cochran-Mantel-Haenszel — P-value from Cochran Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.1736, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.2850, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.3290, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.6938, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1105, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6804, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9704, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6604, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.2447, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4834, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.9189, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4370, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.2894, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.6953, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.4892, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.1954, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.7990, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center

7. Secondary Outcome: Change From Baseline in CGI-S Score at Days 4, 7, 14, 21, 28 and 35
Description: CGI-S is a 7-point scale for assessing the global severity of the participant's illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28 and 35
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -0.1 (0.05) | -0.2 (0.05) | -0.2 (0.07) | -0.2 (0.05)
  Day 7 | -0.3 (0.07) | -0.3 (0.06) | -0.3 (0.10) | -0.3 (0.07)
  Day 14 | -0.6 (0.08) | -0.6 (0.07) | -0.6 (0.11) | -0.5 (0.08)
  Day 21 | -0.6 (0.10) | -0.8 (0.09) | -0.8 (0.13) | -0.7 (0.09)
  Day 28 | -0.7 (0.11) | -0.9 (0.09) | -0.8 (0.14) | -0.8 (0.10)
  Day 35 | -0.9 (0.11) | -1.1 (0.10) | -1.0 (0.14) | -0.8 (0.10)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.4255, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.07 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.9564, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.6363, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.8759, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.9598, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.9789, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.12 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.4671, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.11 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6359, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.11 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.5454, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4188, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.2 to 0.4], Standard Error of Mean 0.13 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5318, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.13 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5683, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.16 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.2972, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.1 to 0.4], Standard Error of Mean 0.14 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4820, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.13 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.9901, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.17 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.6682, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.1111, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.14 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.2400, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.17 — Olanzapine 15 mg BID minus Placebo BID

8. Secondary Outcome: Percentage of Participants Who Are Clinical Global Impression Scale-Improvement (CGI-I) Responders at Days 4, 7, 14, 21, 28, 35 and 42
Description: A CGI-I responder was defined as a participant who had a CGI-I score of 1 (very much improved) or 2 (much improved) at a post-baseline assessment. CGI-I is a 7-point scale for assessing the global improvement of the participant's illness relative to baseline, with ratings from 1=very much improved to 7=very much worse. Missing data were imputed by LOCF.
Time Frame: Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
percentage of participants
  Day 4 (n = 95,108,44,98) | 34.7 (0.27) | 33.3 (0.25) | 43.2 (0.38) | 37.8 (0.27)
  Day 7 (n = 96,111,45,99) | 51.0 (0.30) | 46.8 (0.28) | 60.0 (0.43) | 45.5 (0.30)
  Day 14 (n = 96,111,45,99) | 51.0 (0.31) | 60.4 (0.28) | 71.1 (0.42) | 54.5 (0.30)
  Day 21 (n = 96,111,45,99) | 54.2 (0.32) | 63.1 (0.29) | 75.6 (0.42) | 58.6 (0.31)
  Day 28 (n = 96,111,45,99) | 58.3 (0.36) | 62.2 (0.32) | 73.3 (0.47) | 60.6 (0.35)
  Day 35 (n = 96,111,45,99) | 60.4 (0.34) | 64.0 (0.30) | 82.2 (0.44) | 64.6 (0.32)
  Day 42 (n = 96,111,45,99) | 59.4 (0.40) | 66.7 (0.35) | 84.4 (0.50) | 62.6 (0.38)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.6205, Cochran-Mantel-Haenszel — P-value from Cochran Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.4829, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.3945, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.4076, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.9690, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1170, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.5088, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.3426, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.0762, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5531, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4875, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0692, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.7482, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.8037, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.0859, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.5850, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.9698, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0132, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.7129, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.5074, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0040, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test with an adjustment for pooled center

9. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 7 items of the negative subscale of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS negative subscale score for each participant was sum of the rating assigned to each of the 7 subscale items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -0.7 (0.29) | -0.5 (0.27) | -0.9 (0.42) | -0.8 (0.29)
  Day 7 | -1.2 (0.33) | -1.3 (0.31) | -1.5 (0.47) | -1.1 (0.33)
  Day 14 | -1.6 (0.37) | -2.3 (0.34) | -1.7 (0.51) | -1.8 (0.37)
  Day 21 | -2.3 (0.41) | -2.5 (0.37) | -2.0 (0.56) | -2.3 (0.40)
  Day 28 | -2.5 (0.45) | -3.1 (0.40) | -2.6 (0.59) | -3.0 (0.43)
  Day 35 | -3.3 (0.48) | -3.4 (0.43) | -3.4 (0.63) | -2.6 (0.46)
  Day 42 | -3.3 (0.54) | -4.3 (0.48) | -3.8 (0.68) | -3.2 (0.51)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.8829, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.40 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.5488, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.5 to 1.0], Standard Error of Mean 0.39 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.7830, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.1 to 0.8], Standard Error of Mean 0.50 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.8070, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.0 to 0.8], Standard Error of Mean 0.45 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.5280, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.1 to 0.6], Standard Error of Mean 0.44 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.4025, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.6 to 0.6], Standard Error of Mean 0.57 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6471, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.8 to 1.2], Standard Error of Mean 0.51 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2504, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-1.5 to 0.4], Standard Error of Mean 0.49 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9223, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-1.2 to 1.3], Standard Error of Mean 0.62 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.8839, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-1.0 to 1.2], Standard Error of Mean 0.56 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.8077, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.2 to 0.9], Standard Error of Mean 0.54 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.6216, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-1.0 to 1.7], Standard Error of Mean 0.68 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4248, MMRM — Unadjusted p-value; LS means difference = 0.5, 95% CI 2-sided [-0.7 to 1.7], Standard Error of Mean 0.61 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.7667, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.58 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.6282, MMRM — Unadjusted p-value; LS means difference = 0.4, 95% CI 2-sided [-1.1 to 1.8], Standard Error of Mean 0.72 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.3150, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.9 to 0.6], Standard Error of Mean 0.65 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.1908, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-2.0 to 0.4], Standard Error of Mean 0.61 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.3128, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-2.3 to 0.7], Standard Error of Mean 0.77 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.8812, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.5 to 1.3], Standard Error of Mean 0.73 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.1143, MMRM — Unadjusted p-value; LS means difference = -1.1, 95% CI 2-sided [-2.4 to 0.3], Standard Error of Mean 0.69 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.4418, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-2.3 to 1.0], Standard Error of Mean 0.84 — Olanzapine 15 mg BID minus Placebo BID

10. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 7 items of the positive subscale of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS positive subscale score for each participant was sum of the rating assigned to each of the 7 subscale items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -1.2 (0.29) | -1.6 (0.28) | -2.3 (0.42) | -1.7 (0.30)
  Day 7 | -2.3 (0.39) | -2.8 (0.36) | -3.6 (0.55) | -2.6 (0.38)
  Day 14 | -3.4 (0.45) | -3.9 (0.40) | -4.4 (0.61) | -3.7 (0.43)
  Day 21 | -4.0 (0.52) | -5.0 (0.47) | -5.7 (0.70) | -4.5 (0.51)
  Day 28 | -4.1 (0.59) | -5.7 (0.52) | -6.2 (0.77) | -5.0 (0.56)
  Day 35 | -5.2 (0.60) | -6.3 (0.53) | -6.8 (0.78) | -5.5 (0.57)
  Day 42 | -5.6 (0.65) | -7.2 (0.57) | -7.5 (0.83) | -5.4 (0.61)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.2160, MMRM — Unadjusted p-value; LS means difference = 0.5, 95% CI 2-sided [-0.3 to 1.3], Standard Error of Mean 0.40 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.9494, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.39 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.1834, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.6 to 0.3], Standard Error of Mean 0.50 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.6347, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-0.8 to 1.3], Standard Error of Mean 0.53 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.6917, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.2 to 0.8], Standard Error of Mean 0.51 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1431, MMRM — Unadjusted p-value; LS means difference = -1.0, 95% CI 2-sided [-2.3 to 0.3], Standard Error of Mean 0.66 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.6267, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-0.9 to 1.5], Standard Error of Mean 0.61 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7260, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.3 to 0.9], Standard Error of Mean 0.58 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.3326, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-2.2 to 0.7], Standard Error of Mean 0.74 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4575, MMRM — Unadjusted p-value; LS means difference = 0.5, 95% CI 2-sided [-0.9 to 1.9], Standard Error of Mean 0.72 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4930, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.8 to 0.9], Standard Error of Mean 0.68 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.1886, MMRM — Unadjusted p-value; LS means difference = -1.1, 95% CI 2-sided [-2.8 to 0.6], Standard Error of Mean 0.86 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.2643, MMRM — Unadjusted p-value; LS means difference = 0.9, 95% CI 2-sided [-0.7 to 2.5], Standard Error of Mean 0.80 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.3516, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-2.2 to 0.8], Standard Error of Mean 0.76 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.2068, MMRM — Unadjusted p-value; LS means difference = -1.2, 95% CI 2-sided [-3.1 to 0.7], Standard Error of Mean 0.94 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.7284, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-1.3 to 1.9], Standard Error of Mean 0.82 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.2698, MMRM — Unadjusted p-value; LS means difference = -0.9, 95% CI 2-sided [-2.4 to 0.7], Standard Error of Mean 0.77 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.1510, MMRM — Unadjusted p-value; LS means difference = -1.4, 95% CI 2-sided [-3.3 to 0.5], Standard Error of Mean 0.96 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.8039, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-2.0 to 1.5], Standard Error of Mean 0.88 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0306, MMRM — Unadjusted p-value; LS means difference = -1.8, 95% CI 2-sided [-3.5 to -0.2], Standard Error of Mean 0.83 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0406, MMRM — Unadjusted p-value; LS means difference = -2.1, 95% CI 2-sided [-4.1 to -0.1], Standard Error of Mean 1.03 — Olanzapine 15 mg BID minus Placebo BID

11. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 16 items of the general psychopathology subscale of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS general psychopathology subscale score for each participant was calculated as the sum of the rating assigned to each of the 16 subscale items, and ranged from 16 to 112 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -2.2 (0.49) | -2.7 (0.46) | -2.5 (0.70) | -2.4 (0.49)
  Day 7 | -3.8 (0.69) | -4.9 (0.64) | -4.4 (0.98) | -3.6 (0.68)
  Day 14 | -5.1 (0.73) | -6.2 (0.66) | -6.4 (1.00) | -5.4 (0.71)
  Day 21 | -5.9 (0.84) | -7.4 (0.76) | -7.7 (1.13) | -6.7 (0.81)
  Day 28 | -5.9 (0.93) | -8.2 (0.82) | -8.6 (1.21) | -7.7 (0.88)
  Day 35 | -8.8 (0.88) | -9.2 (0.79) | -10.2 (1.16) | -7.6 (0.84)
  Day 42 | -8.9 (0.97) | -10.1 (0.86) | -10.4 (1.23) | -8.0 (0.92)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.7819, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-1.1 to 1.5], Standard Error of Mean 0.66 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.7030, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.5 to 1.0], Standard Error of Mean 0.65 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.9520, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.7 to 1.6], Standard Error of Mean 0.83 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.7907, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-2.1 to 1.6], Standard Error of Mean 0.95 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1391, MMRM — Unadjusted p-value; LS means difference = -1.4, 95% CI 2-sided [-3.1 to 0.4], Standard Error of Mean 0.91 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.4901, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-3.1 to 1.5], Standard Error of Mean 1.18 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.8079, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-1.7 to 2.2], Standard Error of Mean 1.00 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.3889, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-2.7 to 1.1], Standard Error of Mean 0.95 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.3907, MMRM — Unadjusted p-value; LS means difference = -1.0, 95% CI 2-sided [-3.4 to 1.3], Standard Error of Mean 1.21 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5363, MMRM — Unadjusted p-value; LS means difference = 0.7, 95% CI 2-sided [-1.5 to 3.0], Standard Error of Mean 1.15 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5075, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-2.9 to 1.4], Standard Error of Mean 1.09 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4526, MMRM — Unadjusted p-value; LS means difference = -1.0, 95% CI 2-sided [-3.7 to 1.7], Standard Error of Mean 1.38 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.1548, MMRM — Unadjusted p-value; LS means difference = 1.8, 95% CI 2-sided [-0.7 to 4.3], Standard Error of Mean 1.26 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.6589, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-2.9 to 1.8], Standard Error of Mean 1.19 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.5171, MMRM — Unadjusted p-value; LS means difference = -1.0, 95% CI 2-sided [-3.9 to 2.0], Standard Error of Mean 1.48 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.3133, MMRM — Unadjusted p-value; LS means difference = -1.2, 95% CI 2-sided [-3.6 to 1.2], Standard Error of Mean 1.20 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.1723, MMRM — Unadjusted p-value; LS means difference = -1.6, 95% CI 2-sided [-3.8 to 0.7], Standard Error of Mean 1.13 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0663, MMRM — Unadjusted p-value; LS means difference = -2.6, 95% CI 2-sided [-5.4 to 0.2], Standard Error of Mean 1.42 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.5128, MMRM — Unadjusted p-value; LS means difference = -0.9, 95% CI 2-sided [-3.5 to 1.7], Standard Error of Mean 1.32 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0842, MMRM — Unadjusted p-value; LS means difference = -2.2, 95% CI 2-sided [-4.6 to 0.3], Standard Error of Mean 1.24 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.1217, MMRM — Unadjusted p-value; LS means difference = -2.4, 95% CI 2-sided [-5.4 to 0.6], Standard Error of Mean 1.52 — Olanzapine 15 mg BID minus Placebo BID

12. Secondary Outcome: Change From Baseline in PANSS Marder Factor Positive Symptom Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 8 items of the Marder positive symptom factor of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS Marder factor positive symptom score for each participant was sum of rating assigned to each of the 8 applicable Marder factor items, and ranged from 8 to 56 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -1.3 (0.29) | -1.8 (0.27) | -2.0 (0.41) | -2.0 (0.29)
  Day 7 | -2.5 (0.41) | -2.9 (0.38) | -3.2 (0.58) | -2.8 (0.40)
  Day 14 | -3.9 (0.49) | -4.0 (0.44) | -4.4 (0.67) | -4.1 (0.47)
  Day 21 | -4.5 (0.55) | -5.4 (0.50) | -5.5 (0.74) | -5.1 (0.54)
  Day 28 | -4.8 (0.60) | -6.3 (0.53) | -6.6 (0.78) | -5.6 (0.57)
  Day 35 | -6.1 (0.64) | -6.7 (0.57) | -6.9 (0.84) | -6.1 (0.61)
  Day 42 | -6.8 (0.67) | -7.6 (0.59) | -7.8 (0.86) | -6.2 (0.63)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.0584, MMRM — Unadjusted p-value; LS means difference = 0.7, 95% CI 2-sided [-0.0 to 1.5], Standard Error of Mean 0.39 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.5197, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.5 to 1.0], Standard Error of Mean 0.38 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.9693, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-0.9 to 1.0], Standard Error of Mean 0.49 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.6161, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-0.8 to 1.4], Standard Error of Mean 0.56 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.7880, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.2 to 0.9], Standard Error of Mean 0.54 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.5526, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.8 to 1.0], Standard Error of Mean 0.70 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7647, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-1.1 to 1.5], Standard Error of Mean 0.67 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.8900, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-1.2 to 1.3], Standard Error of Mean 0.64 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7097, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.9 to 1.3], Standard Error of Mean 0.81 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4601, MMRM — Unadjusted p-value; LS means difference = 0.6, 95% CI 2-sided [-0.9 to 2.1], Standard Error of Mean 0.76 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.6288, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.8 to 1.1], Standard Error of Mean 0.72 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.6099, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-2.3 to 1.3], Standard Error of Mean 0.91 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.2790, MMRM — Unadjusted p-value; LS means difference = 0.9, 95% CI 2-sided [-0.7 to 2.5], Standard Error of Mean 0.82 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4253, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-2.1 to 0.9], Standard Error of Mean 0.77 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.3014, MMRM — Unadjusted p-value; LS means difference = -1.0, 95% CI 2-sided [-2.9 to 0.9], Standard Error of Mean 0.96 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.9720, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-1.7 to 1.7], Standard Error of Mean 0.87 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.4758, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-2.2 to 1.0], Standard Error of Mean 0.82 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.4419, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-2.8 to 1.2], Standard Error of Mean 1.03 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.4762, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-2.4 to 1.1], Standard Error of Mean 0.91 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.1046, MMRM — Unadjusted p-value; LS means difference = -1.4, 95% CI 2-sided [-3.1 to 0.3], Standard Error of Mean 0.86 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.1411, MMRM — Unadjusted p-value; LS means difference = -1.6, 95% CI 2-sided [-3.7 to 0.5], Standard Error of Mean 1.06 — Olanzapine 15 mg BID minus Placebo BID

13. Secondary Outcome: Change From Baseline in PANSS Marder Factor Negative Symptom Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 7 items of the Marder negative symptoms factor of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS Marder factor negative symptom score for each participant was sum of the rating assigned to each of the 7 applicable Marder factor items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -1.2 (0.30) | -0.8 (0.28) | -0.8 (0.43) | -0.7 (0.30)
  Day 7 | -1.7 (0.37) | -1.9 (0.34) | -1.8 (0.53) | -1.3 (0.37)
  Day 14 | -2.0 (0.41) | -2.8 (0.37) | -2.2 (0.56) | -2.0 (0.40)
  Day 21 | -2.6 (0.44) | -3.2 (0.40) | -2.6 (0.60) | -2.5 (0.43)
  Day 28 | -2.9 (0.51) | -3.8 (0.45) | -3.2 (0.67) | -3.5 (0.49)
  Day 35 | -3.5 (0.52) | -3.9 (0.46) | -4.1 (0.68) | -3.0 (0.49)
  Day 42 | -3.4 (0.53) | -4.7 (0.47) | -4.3 (0.67) | -4.0 (0.51)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.2754, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.2 to 0.4], Standard Error of Mean 0.40 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.8500, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-0.8 to 0.7], Standard Error of Mean 0.39 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.8439, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.1 to 0.9], Standard Error of Mean 0.51 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.4741, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.4 to 0.6], Standard Error of Mean 0.51 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.2158, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-1.6 to 0.4], Standard Error of Mean 0.49 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.5060, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.7 to 0.8], Standard Error of Mean 0.63 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9956, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-1.1 to 1.1], Standard Error of Mean 0.56 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.1624, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.8 to 0.3], Standard Error of Mean 0.53 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7662, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.5 to 1.1], Standard Error of Mean 0.68 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.8363, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.3 to 1.1], Standard Error of Mean 0.61 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.2388, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.8 to 0.5], Standard Error of Mean 0.58 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.9435, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.5 to 1.4], Standard Error of Mean 0.73 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4267, MMRM — Unadjusted p-value; LS means difference = 0.6, 95% CI 2-sided [-0.8 to 1.9], Standard Error of Mean 0.70 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.6810, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.6 to 1.0], Standard Error of Mean 0.65 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.7673, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-1.4 to 1.9], Standard Error of Mean 0.82 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.4830, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.9 to 0.9], Standard Error of Mean 0.70 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.2128, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-2.1 to 0.5], Standard Error of Mean 0.66 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.1756, MMRM — Unadjusted p-value; LS means difference = -1.1, 95% CI 2-sided [-2.8 to 0.5], Standard Error of Mean 0.83 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.4246, MMRM — Unadjusted p-value; LS means difference = 0.6, 95% CI 2-sided [-0.8 to 2.0], Standard Error of Mean 0.72 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.2873, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-2.1 to 0.6], Standard Error of Mean 0.68 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.7308, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.9 to 1.4], Standard Error of Mean 0.83 — Olanzapine 15 mg BID minus Placebo BID

14. Secondary Outcome: Change From Baseline in PANSS Marder Factor Disorganized Thought Symptom Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 7 items of the Marder disorganized thoughts factor of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS Marder factor disorganized thought symptom score for each participant was sum of rating assigned to each of the 7 applicable Marder factor items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -0.3 (0.24) | -0.7 (0.22) | -1.1 (0.34) | -0.7 (0.24)
  Day 7 | -1.0 (0.32) | -1.4 (0.29) | -1.6 (0.45) | -0.7 (0.31)
  Day 14 | -1.3 (0.36) | -2.0 (0.33) | -2.2 (0.49) | -1.5 (0.35)
  Day 21 | -2.3 (0.41) | -2.5 (0.37) | -2.7 (0.54) | -2.1 (0.39)
  Day 28 | -2.4 (0.42) | -3.1 (0.37) | -3.1 (0.54) | -2.4 (0.40)
  Day 35 | -3.5 (0.43) | -3.5 (0.38) | -4.3 (0.56) | -2.4 (0.41)
  Day 42 | -3.8 (0.45) | -4.3 (0.40) | -4.7 (0.58) | -2.7 (0.43)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.2116, MMRM — Unadjusted p-value; LS means difference = 0.4, 95% CI 2-sided [-0.2 to 1.0], Standard Error of Mean 0.32 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.9039, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-0.6 to 0.7], Standard Error of Mean 0.31 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.2959, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.2 to 0.4], Standard Error of Mean 0.4 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.5909, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.1 to 0.6], Standard Error of Mean 0.44 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1489, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-1.4 to 0.2], Standard Error of Mean 0.42 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.1000, MMRM — Unadjusted p-value; LS means difference = -0.9, 95% CI 2-sided [-2.0 to 0.2], Standard Error of Mean 0.54 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7830, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.8 to 1.1], Standard Error of Mean 0.49 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2679, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.4 to 0.4], Standard Error of Mean 0.47 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2321, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.9 to 0.5], Standard Error of Mean 0.60 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.7368, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.3 to 0.9], Standard Error of Mean 0.56 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.4606, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.4 to 0.7], Standard Error of Mean 0.53 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.3241, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-2.0 to 0.7], Standard Error of Mean 0.66 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.9860, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-1.1 to 1.1], Standard Error of Mean 0.57 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.1890, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.8 to 0.3], Standard Error of Mean 0.53 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.3030, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-2.0 to 0.6], Standard Error of Mean 0.67 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0550, MMRM — Unadjusted p-value; LS means difference = -1.1, 95% CI 2-sided [-2.3 to 0.0], Standard Error of Mean 0.58 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0415, MMRM — Unadjusted p-value; LS means difference = -1.1, 95% CI 2-sided [-2.2 to -0.0], Standard Error of Mean 0.55 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.0058, MMRM — Unadjusted p-value; LS means difference = -1.9, 95% CI 2-sided [-3.3 to -0.6], Standard Error of Mean 0.69 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0691, MMRM — Unadjusted p-value; LS means difference = -1.1, 95% CI 2-sided [-2.3 to 0.1], Standard Error of Mean 0.62 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0063, MMRM — Unadjusted p-value; LS means difference = -1.6, 95% CI 2-sided [-2.7 to -0.5], Standard Error of Mean 0.58 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.0056, MMRM — Unadjusted p-value; LS means difference = -2.0, 95% CI 2-sided [-3.4 to -0.6], Standard Error of Mean 0.71 — Olanzapine 15 mg BID minus Placebo BID

15. Secondary Outcome: Change From Baseline in PANSS Marder Factor Hostility/Excitement Symptom Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 4 items of the Marder hostility/excitement factor of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS Marder factor hostility/excitement symptom score for each participant was sum of rating assigned to each of the 4 applicable Marder factor items, and ranged from 4 to 28 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -0.4 (0.25) | -0.3 (0.23) | -0.7 (0.36) | -0.5 (0.25)
  Day 7 | -0.5 (0.28) | -0.5 (0.26) | -1.0 (0.40) | -0.7 (0.28)
  Day 14 | -0.9 (0.30) | -0.8 (0.27) | -1.2 (0.41) | -0.9 (0.30)
  Day 21 | -0.8 (0.33) | -0.9 (0.30) | -1.8 (0.44) | -1.0 (0.32)
  Day 28 | -0.5 (0.41) | -0.8 (0.36) | -1.6 (0.53) | -1.0 (0.39)
  Day 35 | -1.4 (0.37) | -1.5 (0.32) | -2.0 (0.47) | -1.4 (0.35)
  Day 42 | -1.1 (0.41) | -1.8 (0.36) | -1.9 (0.52) | -1.1 (0.39)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.7847, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.6 to 0.8], Standard Error of Mean 0.34 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.5859, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.5 to 0.8], Standard Error of Mean 0.33 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.6413, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.43 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.7307, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.38 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.7176, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.37 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.4860, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.3 to 0.6], Standard Error of Mean 0.48 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.9321, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.41 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.7691, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.7 to 0.9], Standard Error of Mean 0.39 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.5694, MMRM — Unadjusted p-value; LS means difference = -0.3, 95% CI 2-sided [-1.3 to 0.7], Standard Error of Mean 0.50 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5583, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-0.6 to 1.2], Standard Error of Mean 0.45 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.7307, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.7 to 1.0], Standard Error of Mean 0.43 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.1715, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.8 to 0.3], Standard Error of Mean 0.54 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.4219, MMRM — Unadjusted p-value; LS means difference = 0.4, 95% CI 2-sided [-0.6 to 1.5], Standard Error of Mean 0.55 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.7437, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.9 to 1.2], Standard Error of Mean 0.52 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.3110, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.9 to 0.6], Standard Error of Mean 0.65 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.9805, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-1.0 to 1.0], Standard Error of Mean 0.50 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.8741, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.0 to 0.8], Standard Error of Mean 0.47 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.3288, MMRM — Unadjusted p-value; LS means difference = -0.6, 95% CI 2-sided [-1.7 to 0.6], Standard Error of Mean 0.58 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.9336, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-1.0 to 1.1], Standard Error of Mean 0.56 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.1722, MMRM — Unadjusted p-value; LS means difference = -0.7, 95% CI 2-sided [-1.7 to 0.3], Standard Error of Mean 0.52 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.1909, MMRM — Unadjusted p-value; LS means difference = -0.8, 95% CI 2-sided [-2.1 to 0.4], Standard Error of Mean 0.64 — Olanzapine 15 mg BID minus Placebo BID

16. Secondary Outcome: Change From Baseline in PANSS Marder Factor Anxiety/Depression Symptom Score at Days 4, 7, 14, 21, 28, 35 and 42
Description: This measure reports results for the 4 items of the Marder anxiety/depression factor of the PANSS, which is a 30-item clinician-rated instrument used to assess schizophrenia symptoms. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. PANSS Marder factor anxiety/depression symptom score for each participant was sum of rating assigned to each of the 4 applicable Marder factor items, and ranged from 4 to 28 with a higher score indicating greater severity of symptoms. Measure reports change from baseline; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Days 4, 7, 14, 21, 28, 35 and 42
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Number analyzed (Participants) | 96 | 111 | 45 | 99
score on a scale
  Day 4 | -0.9 (0.27) | -1.2 (0.25) | -1.0 (0.38) | -0.9 (0.27)
  Day 7 | -1.5 (0.30) | -2.2 (0.28) | -1.8 (0.43) | -1.7 (0.30)
  Day 14 | -1.9 (0.31) | -2.9 (0.28) | -2.5 (0.42) | -2.5 (0.30)
  Day 21 | -2.1 (0.32) | -3.0 (0.29) | -2.7 (0.42) | -3.1 (0.31)
  Day 28 | -1.9 (0.36) | -3.2 (0.32) | -2.8 (0.47) | -3.4 (0.35)
  Day 35 | -3.0 (0.34) | -3.6 (0.30) | -3.2 (0.44) | -3.2 (0.32)
  Day 42 | -2.9 (0.40) | -3.4 (0.35) | -3.1 (0.50) | -3.0 (0.38)
Statistical Analysis 1: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.9851, MMRM — Unadjusted p-value; LS means difference = 0.0, 95% CI 2-sided [-0.7 to 0.7], Standard Error of Mean 0.37 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 2: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.4912, MMRM — Unadjusted p-value; LS means difference = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.36 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 3: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 4; Test type: Superiority or Other; p = 0.8559, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.0 to 0.8], Standard Error of Mean 0.46 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 4: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.5635, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.6 to 1.1], Standard Error of Mean 0.41 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 5: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.2321, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.3 to 0.3], Standard Error of Mean 0.40 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 6: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 7; Test type: Superiority or Other; p = 0.8867, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.1 to 0.9], Standard Error of Mean 0.52 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 7: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.1499, MMRM — Unadjusted p-value; LS means difference = 0.6, 95% CI 2-sided [-0.2 to 1.4], Standard Error of Mean 0.42 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 8: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.2860, MMRM — Unadjusted p-value; LS means difference = -0.4, 95% CI 2-sided [-1.2 to 0.4], Standard Error of Mean 0.40 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 9: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 14; Test type: Superiority or Other; p = 0.8978, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.1 to 0.9], Standard Error of Mean 0.51 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 10: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.0283, MMRM — Unadjusted p-value; LS means difference = 1.0, 95% CI 2-sided [0.1 to 1.8], Standard Error of Mean 0.44 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 11: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.8667, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-0.7 to 0.9], Standard Error of Mean 0.41 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 12: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 21; Test type: Superiority or Other; p = 0.5044, MMRM — Unadjusted p-value; LS means difference = 0.3, 95% CI 2-sided [-0.7 to 1.4], Standard Error of Mean 0.52 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 13: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.0040, MMRM — Unadjusted p-value; LS means difference = 1.4, 95% CI 2-sided [0.5 to 2.4], Standard Error of Mean 0.49 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 14: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.6330, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.7 to 1.1], Standard Error of Mean 0.46 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 15: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 28; Test type: Superiority or Other; p = 0.2981, MMRM — Unadjusted p-value; LS means difference = 0.6, 95% CI 2-sided [-0.5 to 1.7], Standard Error of Mean 0.57 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 16: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.6556, MMRM — Unadjusted p-value; LS means difference = 0.2, 95% CI 2-sided [-0.7 to 1.1], Standard Error of Mean 0.45 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 17: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.2889, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.3 to 0.4], Standard Error of Mean 0.43 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 18: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 35; Test type: Superiority or Other; p = 0.9399, MMRM — Unadjusted p-value; LS means difference = -0.0, 95% CI 2-sided [-1.1 to 1.0], Standard Error of Mean 0.53 — Olanzapine 15 mg BID minus Placebo BID
Statistical Analysis 19: Comparison: Asenapine 2.5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.8955, MMRM — Unadjusted p-value; LS means difference = 0.1, 95% CI 2-sided [-1.0 to 1.1], Standard Error of Mean 0.54 — Asenapine 2.5 mg BID minus Placebo BID
Statistical Analysis 20: Comparison: Asenapine 5 mg BID vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.3681, MMRM — Unadjusted p-value; LS means difference = -0.5, 95% CI 2-sided [-1.5 to 0.5], Standard Error of Mean 0.51 — Asenapine 5 mg BID minus Placebo BID
Statistical Analysis 21: Comparison: Olanzapine 15 mg QD vs Placebo BID; Day 42; Test type: Superiority or Other; p = 0.8215, MMRM — Unadjusted p-value; LS means difference = -0.1, 95% CI 2-sided [-1.4 to 1.1], Standard Error of Mean 0.62 — Olanzapine 15 mg BID minus Placebo BID

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 10 weeks)
Arm/Group | Asenapine 2.5 mg BID | Asenapine 5 mg BID | Olanzapine 15 mg QD | Placebo BID
Serious Adverse Events (participants affected / at risk) | 5/97 | 5/113 | 1/46 | 8/101
Other Adverse Events (participants affected / at risk) | 27/97 | 47/113 | 17/46 | 29/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 2.5 mg BID (N=97) | Asenapine 5 mg BID (N=113) | Olanzapine 15 mg QD (N=46) | Placebo BID (N=101)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Schizophrenia, paranoid type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 2.5 mg BID (N=97) | Asenapine 5 mg BID (N=113) | Olanzapine 15 mg QD (N=46) | Placebo BID (N=101)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 4 (4) | 7 (7) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (12) | 10 (10) | 4 (6) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3) | 7 (7) | 5 (5) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 7 (8) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 7 (10) | 8 (9) | 4 (5) | 12 (13)
Insomnia (Psychiatric disorders) | 9 (9) | 17 (21) | 4 (4) | 14 (20)
Schizophrenia (Psychiatric disorders) | 6 (6) | 4 (4) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is planned to first publish/present trial results together with the other sites, unless permission is obtained from Sponsor to publish separate results. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. If there is disagreement concerning appropriateness of the materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve disagreement prior to submission for publication.